CLINICAL TRIAL: NCT04016012
Title: Overweight and Obesity in Relation to Type II Melitus,Diabetes A Randomised Controlled Trial
Brief Title: Overweight and Obesity in Relation to Type ll Diabetes Melitus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mukuba University (Other)
Collaborators: University of Zambia (Other); Afe Babalola University, Nigeria (Unknown); Buea University, Cameroon (Unknown); Sokoine University of Agriculture (Other); Kitwe Teaching Hospital, Zambia (Unknown); National Science and Technology Council (U.S. Federal Agency)
Responsible Party: Principal Investigator, Given Chipili, Dr, Mukuba University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MU0619
Record Dates: First submitted 2019-07-07; First posted 2019-07-11 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Diabetes Mellitus, Type 2; Overweight and Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: The intervention group will receive a diabetic controlled diet using local Zambian foods for 8 weeks and standard health care for 8 weeks while the control group will eat their usual food in their home and receive standard health care for eight (8) weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): Participants in the intervention group will receive local zambian foods and standard health care for eight (8) weeks.
  Interventions: Dietary Supplement: Local Zambian Foods
- Control arm (No Intervention): The control group will have their usual (standard) diet in their home and receive standard health care for eight (8) weeks.

INTERVENTIONS:
Dietary Supplement: Local Zambian Foods — Each week, participants in the intervention group will collect a pack of foodstuffs to last a week from the research site. The packs will be adjusted according to the weight of the participant and daily recommended allowances. Packaging of foodstuffs will be done in the food service lab at the Mukuba University. Instructions on how to prepare and use the food will be given to the participants. All food Items will be labelled diabetic food to avoid intra-household sharing.
  Arms: Intervention arm

SUMMARY:
The aim of the study is to evaluate the efficacy of local Zambian food in improving metabolic profiles of overweight/obese type ll diabetic patients in Kitwe district

ELIGIBILITY:
Inclusion Criteria:

* Diabetic patients attending Kitwe Teaching Hospital
* 18 years and above
* Body Mass Index of 25 and above
* Willing to follow the diet plan and eat food provided
* Not enrolled in other clinical studies

Exclusion Criteria:

* Eating disorder or any psychosocial or scheduling factors that could impede study outcomes
* Have renal or liver problem
* Pregnant women
* Breast feeding women
* HIV positive individuals

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-04-30 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-10-15 (Estimated)

PRIMARY OUTCOMES:
Change in Blood glucose levels | At baseline and 8 weeks
  Fingertip blood sugar test using: blood glucose meter, test strips, lancet device, dry swabs, methylated spirit and a sharps box.

SECONDARY OUTCOMES:
Change in Body weight | At baseline and 8 weeks
  Weight will be measured using the Seca adult scale
Change of Body Mass Index (BMI) | At baseline and 8 weeks
  Hand held BMI machine will be used to determine the BMI of each participant.

CONTACTS AND LOCATIONS:
Overall Officials: Given Chipili, Principal Investigator — Mukuba University, Kitwe, Zambia
Locations (1):
- Kitwe Teaching Hospital, Kitwe, Copperbelt, Zambia

IPD SHARING:
Plan to Share IPD: Yes
Data collected in this study will be published online
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 6 months after the study ends.
Access Criteria: Mukuba University Website
URL: http://www.mukuba.edu.zm